CLINICAL TRIAL: NCT01431300
Title: Dose-varied Evaluation of Ablavar-enhanced MR Angiography of the Central Veins of the Chest in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Pro00022334; CG 10011 (Other Grant/Funding Number: Lantheus Medical Imaging)
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: central veins; thorax; superior vena cava; Central vein imaging
MeSH Terms: interventions — gadofosveset trisodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.03 mmol/kg (Active Comparator): FDA-approved dose for lower extremity arterial imaging
  Interventions: Drug: gadofosveset
- 0.02 mmol/kg (Experimental)
  Interventions: Drug: gadofosveset
- 0.01 mmol/kg (Experimental)
  Interventions: Drug: gadofosveset

INTERVENTIONS:
Drug: gadofosveset — Intravenous administration of the specified dosage of gadolinium contrast agent
  Other Names: Ablavar

SUMMARY:
The purpose of this study is to assess the image quality of Ablavar-enhanced MR angiography of the central veins of the chest, and to determine whether dose reduction can be performed while maintaining image quality. This will be a prospective randomized study, in which healthy volunteers will be recruited to undergo a central veins magnetic resonance angiogram (MRA). They will receive either the FDA-approved dose or a lower dose of Ablavar. Quantitative and qualitative analysis will be performed on the images.

ELIGIBILITY:
Inclusion Criteria:

* healthy male or female subjects between 18-45 years of age

Exclusion Criteria:

* Pregnant and lactating females
* known renal impairment
* allergy to gadolinium-based contrast
* metallic implanted devices
* claustrophobia.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Y Kim, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Kim CY, Heye T, Bashir MR, Gebhard TA, Merkle EM. Gadofosveset-enhanced magnetic resonance angiography of the thoracic vasculature in the equilibrium phase: feasibility and impact of dose. J Comput Assist Tomogr. 2013 Sep-Oct;37(5):732-6. doi: 10.1097/RCT.0b013e318299dde9. PMID 24045249

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.01 mmol/kg of Gadofosveset; 0.02 mmol/kg of Gadofosveset: Intravenous administration of gadofosveset via power injector at onset of MRI image acquisition
- 0.03 mmol/kg of Gadofosveset: Intravenous administration of gadofosveset via power injector at onset of MRI image acquisition. This is the FDA-approved dose for lower extremity arterial imaging
Period: Overall Study
Arm/Group | 0.01 mmol/kg of Gadofosveset | 0.02 mmol/kg of Gadofosveset | 0.03 mmol/kg of Gadofosveset
Started | 11 (One subject with indeterminate pregnancy test, subject declined to proceed) | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 0.01 mmol/kg; 0.02 mmol/kg: gadofosveset : Intravenous administration of the specified dosage of gadolinium contrast agent
- 0.03 mmol/kg: FDA-approved dose for lower extremity arterial imaging
  gadofosveset : Intravenous administration of the specified dosage of gadolinium contrast agent
- Total: Total of all reporting groups
Arm/Group | 0.01 mmol/kg | 0.02 mmol/kg | 0.03 mmol/kg | Total
Number analyzed (Participants) | 11 | 10 | 10 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 10 | 31
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 22.2 (5.3) | 24.6 (8.1) | 24.1 (7.5) | 23.4 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 1 | 8
  Male | 10 | 4 | 9 | 23

OUTCOME MEASURES:

1. Primary Outcome: Imaging Quality Score
Description: Two radiologists assessed imaging quality of each central venous segment for each patient, in order to compare imaging quality between each of the three doses administered. The visualization score for each venous segments was as follows:
  1. poor / nondiagnostic
  2. adequate
  3. good
  4. excellent
Time Frame: 14 weeks
Measure: Mean (Full Range); unit: Units on a visualization score scale
Arm/Group | 0.01 mmol/kg | 0.02 mmol/kg | 0.03 mmol/kg
Number analyzed (Participants) | 10 | 10 | 10
Units on a visualization score scale | 2.1 [1 to 4] | 2.1 [1 to 4] | 2.3 [1 to 4]

2. Secondary Outcome: Quantitative Analysis Noise Ratios
Description: Signal-to-noise and contrast-to-noise ratios were calculated for each central venous segment, to determine the magnitude of difference in each of the three administered doses. The ratio's were calculated as follows:
  Signal-to-noise ratio: signal intensity of vessel segment / standard deviation of signal intensity of the background.
  Contrast-to-noise ratio = (signal intensity of vessel segment minus signal intensity of adjacent muscle) / standard deviation of signal intensity of the background.
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 0.01 mmol/kg | 0.02 mmol/kg | 0.03 mmol/kg
Number analyzed (Participants) | 10 | 10 | 10
ratio
  signal to noise ratio | 81 (17) | 119 (28) | 135 (25)
  contrast to noise ratio | 37 (14) | 60 (28) | 80 (25)
Statistical Analysis 1: Comparison: 0.01 mmol/kg vs 0.03 mmol/kg; signal-to-noise (SNR) ratios of the central veins in the 0.01 mmol/kg and 0.03mmol/kg dose groups were compared; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 54, Standard Deviation 12
Statistical Analysis 2: Comparison: 0.01 mmol/kg vs 0.03 mmol/kg; contrast-to-noise (CNR) ratios of the central veins in the 0.01 mmol/kg and 0.03mmol/kg dose groups were compared; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 43, Standard Deviation 19

ADVERSE EVENTS:
Arm/Group | 0.01 mmol/kg | 0.02 mmol/kg | 0.03 mmol/kg
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No